CLINICAL TRIAL: NCT02033447
Title: Magnetic Nanoparticle Thermoablation-Retention and Maintenance in the Prostate:A Phase 0 Study in Men
Acronym: MAGNABLATE I
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University College London Hospitals (Other)
Responsible Party: Principal Investigator, Hashim Uddin Ahmed, MRC Clinician Scientist, University College London Hospitals
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 13/0257; National Institute for Health (Other Grant/Funding Number: II-SB-0712-20001)
Record Dates: First submitted 2014-01-06; First posted 2014-01-10 (Estimated); Last update posted 2017-05-10 (Actual); Status verified 2017-05

CONDITIONS: Prostate Cancer
Keywords: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Magnetic Nanoparticle Injection (Experimental): Patients undergoing radical cystoprostatectomy or prostatectomy
  Interventions: Other: Magnetic Nanoparticle Injection

INTERVENTIONS:
Other: Magnetic Nanoparticle Injection

SUMMARY:
Men with early prostate cancer face a number of options which lie at the extremes of care. On one hand, active surveillance involves monitoring the disease and on the other, immediate treatment involves surgery or radiotherapy. The difference between these two strategies in terms of reducing the chance of a man dying from his disease is small. Not only is the benefit small, surgery or radiotherapy carry significant side-effects. These occur because of damage to surrounding tissue resulting in incontinence of urine (1 in 5), erectile dysfunction (1 in 2) and back-passage bleeding, diarrhoea or discomfort (1 in 10).

The investigators have been working on new forms of treatment that use heat, light or cold to destroy tissue and minimise treatment-related harms. The investigators have not yet found one that delivers the ideal treatment. The ideal treatment is one that can be done under local anaesthetic, can effectively destroy areas of cancer, limit damage to surrounding tissues, is repeatable, and adaptable to future discoveries such as molecular targeting of cancer cells.

The investigators think magnetic thermoablation may be able to deliver on these ideal attributes. Magnetic thermoablation involves injecting magnetic iron nanoparticles directly into the cancer. When a magnetic field is applied close to them, these nanoparticles heat up to very high temperatures that kill cells. Magnetic thermoablation does not use x-rays or surgical incisions. The investigators have done a lot of the preclinical work already to develop this type of treatment. The investigators now need to develop a system that can be used to treat prostate cancer. However, before the investigators can do this, they need to test whether the magnetic nanoparticles actually stay where they are injected. The consequences of them moving to areas that they should not can be serious. First, the nanoparticles could move away from the cancer which means the cancer will not be heated effectively. Second, the nanoparticles could move to sensitive structures around the prostate (back-passage, bladder, sphincter muscle controlling urine flow, nerves controlling erections). If this happens, damage of those sensitive structures could occur leading to side-effects.

The investigators propose a study to try and find out what happens to those nanoparticles. The study will involve approaching men who are having their prostates removed by radical surgery. If these patients agree to participate, the investigators will inject their prostate with varying amounts of nanoparticles. The investigators will NOT heat them up. The investigators will use special scans and, once they have had their surgery, to look at the pathology specimens to see where the nanoparticles have gone. The actual nanoparticles are not harmful but the process of injection can carry a small amount of harm. If the nanoparticles stay where they are injected, the investigators will then be able to run another study in which we treat men who have prostate cancer with magnetic thermoablation.

DETAILED DESCRIPTION:
PRIMARY

1.1 To conduct a dose escalation safety trial of magnetic nanoparticles injected into the prostates of men prior to cystoprostatectomy. 1.2 To conduct a dose escalation safety trial of magnetic nanoparticles injected into the prostates of men prior to prostatectomy. 1.3 To evaluate ex-vivo prostates with a special marker to determine the retention and distribution of the magnetic nanoparticles in relation to the intended target area at time of injection

SECONDARY 2.1 To evaluate the anatomical distribution of magnetic nanoparticles compared with injection site in prostate assessed by both Perls' staining and postoperative imaging (MRI and CT) of the ex vivo tissue

ELIGIBILITY:
Inclusion Criteria:

1. Patients undergoing radical cystoprostatectomy for bladder cancer
2. Patients undergoing radical prostatectomy for prostate cancer
3. Patients giving informed consent

Exclusion Criteria:

1. Have taken any form of hormones (except 5-alpha reductase inhibitors) within the last 6 months
2. Unable to have MRI scan or CT scan, or in whom artefact would reduce scan quality
3. Unable to have general or regional anaesthesia
4. Patients on immunosuppression or predefined immunosuppressed state
5. Patients with a coagulopathy predisposing to bleeding to clot formation
6. Patients with an inherited or acquired condition limiting metabolism of iron
7. Unable to give informed consent

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2013-12; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Adverse Events as a Measure of Safety and Tolerability | outcome measures assessed every month and presented at 12 months for the primary end points
  1.1 dose escalation safety trial of magnetic nanoparticles injected into the prostates of patients prior to cystoprostatectomy.
  1.2 a dose escalation safety trial of magnetic nanoparticles injected into the prostates of patients prior to prostatectomy.
  1.3 ex-vivo prostates with a special marker to determine the retention and distribution of the magnetic nanoparticles in relation to the intended target area at time of injection

SECONDARY OUTCOMES:
The anatomical distribution of magnetic nanoparticles | every month will be assessed and presented at 12 months for the secondary end points
  2.1 anatomical distribution of magnetic nanoparticles compared with injection site in prostate assessed by both Perls' staining and postoperative imaging (MRIand CT) of the ex vivo tissue

CONTACTS AND LOCATIONS:
Overall Officials: Hashim Ahmed, MbChB, PhD, Principal Investigator — MRC Clinical Scientist
Locations (1):
- University College London Hospital, London, United Kingdom